CLINICAL TRIAL: NCT03629106
Title: Effects of Extended Cannabis Abstinence on Clinical and Cognitive Outcomes in Patients With Co-Morbid Bipolar Disorder and Cannabis Use Disorder
Brief Title: Effects of Cannabis Abstinence on Symptomology and Cognition in Bipolar Disorder
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of funding
Sponsor: Centre for Addiction and Mental Health (Other)
Responsible Party: Principal Investigator, Tony George, Chief, Addictions Division, Centre for Addiction and Mental Health
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 053/2018
Record Dates: First submitted 2018-08-09; First posted 2018-08-14 (Actual); Last update posted 2023-09-11 (Actual); Status verified 2023-09

CONDITIONS: Cannabis Use Disorder; Bipolar Disorder; Cognition
Keywords: Bipolar Disorder; Cannabis Use Disorder; Cognitive Function
MeSH Terms: conditions — Bipolar Disorder

STUDY DESIGN:
Intervention Model Description: Randomized open-label trial to compare two arms: 1) contingent reinforcement and 2) non-contingent reinforcement.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Contingent Reinforcement (Experimental): The Contingent Reinforcement (CR) group (n=26) will be given an abstinence bonus at the successful completion of a 28-Day cannabis abstinence verified by self-report and urinary THC-COOH level <20 ng/ml.
  Interventions: Behavioral: Weekly Behavioral Coaching Session
- No Contingent Reinforcement (Experimental): The Non-Contingent Reinforcement (NCR) group (n=26) will not be given an abstinence bonus at the successful completion of a 28-Day cannabis abstinence.
  Interventions: Behavioral: Weekly Behavioral Coaching Session

INTERVENTIONS:
Behavioral: Weekly Behavioral Coaching Session — The participants will be provided with a 20-minute individual behavioral support session weekly for 4 weeks (28 days abstinence), designed to provide them with tools and techniques to manage the craving and withdrawal symptoms that occur with cessation.

SUMMARY:
The objective of this study is to assess the changes in symptoms and cognition that occur after a 28-day abstinence period in patients with comorbid Cannabis Use Disorder (CUD) and Bipolar (Type I or II) disorder. Stabilized bipolar patients (N=52) with CUD will be randomly assigned to one of two groups: 1) A contingent reinforcement (CR) group (n=26); 2) a non-contingent reinforcement (NCR) group (n=26). The study will include a total of 8 visits to the CAMH Russell site (screening, training, baselines, week 1-4, follow-up). Participants should be between the ages of 18-60, meet criteria for CUD (moderate to severe), meet criteria for Bipolar Disorder, be on a stable dose of mood stabilizing medication(s), and be non-treatment seeking cannabis user. The visits will take up a total of approximately 22.5 hours with compensation for time provided for both groups. These visits will involve multiple clinical, substance use, and cognitive assessments. Abstinence will be maintained by weekly behavioural coaching sessions and contingency reinforcement for the CR group.

ELIGIBILITY:
Inclusion Criteria:

* All participants must be between the ages 18-60
* Meet SCID for DSM-5 diagnostic criteria for cannabis use disorder, moderate to severe
* Meet SCID for DSM-5 diagnostic criteria for Bipolar Disorder (Type I or II)
* Be an outpatient receiving a stable dose of mood stabilizing medication(s) for at least one month
* Have a Hamilton Depression Rating Scale (HDRS-17) baseline assessment in the range of 12-25
* Have a Full-Scale IQ of at least 80 as determined by the WTAR
* Be a non-treatment seeking cannabis user
* Evidence of sufficient motivation and effort as measured by a Test of Memory Malingering (TOMM) score of at least 45
* Y-MRS baseline score in the range of 0-15

Exclusion Criteria:

* Meets criteria for abuse or dependence of alcohol or other illicit substances within the past 6 months (with the exception of cannabis, nicotine, or caffeine)
* Positive urine screen for illicit substances other than cannabis, nicotine, or caffeine
* Current suicidal or homicidal ideation
* Psychotic disorder diagnosis (e.g. schizoaffective disorder, major depression with psychotic features) as determined by the SCID
* Treatment seeking for cannabis use
* Head Injury > 5 minutes LOC
* Exceed upper and lower cut-offs on HSRD-17 and YMRS

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2022-08-31 (Estimated); Study Completion 2022-08-31 (Estimated)

PRIMARY OUTCOMES:
The effects of 28 day cannabis abstinence on change in depressive symptoms in cannabis-dependent patients with bipolar disorder as assessed by the Hamilton Rating Scale for Depression (HRSD). | Weekly (Day 0, Day 7, Day 14, Day 21, Day 28) and at 8 weeks (Follow-up Day 56)
  The clinical assessment will be administered weekly during the abstinence period and conducted by study personnel.
The effects of 28 day cannabis abstinence on change in hypomania symptoms in cannabis-dependent patients with bipolar disorder as assessed by the Young Mania Rating Scale (YMRS). | Weekly (Day 0, Day 7, Day 14, Day 21, Day 28) and at 8 weeks (Follow-up Day 56)
  The clinical assessment will be administered weekly during the abstinence period and conducted by study personnel.

SECONDARY OUTCOMES:
The effects of 28 day cannabis abstinence on change in cognitive function in cannabis dependent patients with bipolar disorder as assessed by a cognitive battery administered at Baseline, Week 2, Endpoint and Follow-Up. | Bi-Weekly (Day 0, Day 14, Day 28) and at 8 Weeks (Follow-up Day 56)
  The cognitive battery will include the primary outcome of motivation and effort (assessed by TOMM) and will be compared to baseline (Day 1) performance. Cortical inhibition will also be assessed and compared.
The effects of 28 day cannabis abstinence on change in co-occurring anxiety in cannabis dependent patients with bipolar disorder as assessed by the Beck Anxiety Inventory (BAI). | Weekly (Day 0, Day 7, Day 14, Day 21, Day 28) and at 8 weeks (Follow-up Day 56)
  The clinical assessment will be administered at Baseline, weekly during the abstinence period and Follow-up and will be conducted by study personnel.

CONTACTS AND LOCATIONS:
Overall Officials: Tony George, M.D., FRCPC, Principal Investigator — Centre for Addiction and Mental Health
Locations (1):
- Centre for Addiction and Mental Health, Toronto, Ontario, Canada